CLINICAL TRIAL: NCT07391397
Title: Reducing Rural Health Disparities by Empowering People to Minimize PFAS Exposure and Improve Cardiovascular Health
Brief Title: Assessing PFAS Exposure (APEX) for Better Health
Acronym: APEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Million Marker Wellness, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Renown Health (Other)
Responsible Party: Principal Investigator, Jenna Hua, Environmental Health Scientist, Million Marker Wellness, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2331153; 1R43HL179154-01A1 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Environmental Health Effects
Keywords: PFAS; Environmental Health; EDCs
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other): All participants who take the PFAS Blood Test
  Interventions: Behavioral: Blood Test and Report Back

INTERVENTIONS:
Behavioral: Blood Test and Report Back — Participants take an at home blood test to test their PFAS levels and receive a report back with recommendations to reduce exposures.

SUMMARY:
The goal of this observational study is to determine whether a personalized PFAS (per- and polyfluoroalkyl substances) blood test and educational report-back can improve environmental health literacy (EHL), empower exposure reduction behaviors, and promote cardiovascular wellness among rural adults. The main questions it aims to answer are: Does receiving a personalized PFAS test result and educational report-back increase environmental health literacy among rural participants and healthcare providers? Does increased EHL lead to greater readiness and actions to reduce PFAS exposure and improve wellness outcomes (e.g., reduced stress, improved sleep, increased sense of control) Researchers will compare changes from pre- to post-intervention among participants who receive the personalized PFAS report-back to see if there are measurable improvements in knowledge, behavior, and wellbeing. Participants will: Provide a mail-in blood spot sample for PFAS testing using a validated laboratory method (Relentless Health). Complete online surveys before and after receiving results to assess PFAS knowledge, exposure behaviors, and wellness outcomes. Receive a personalized PFAS report-back summarizing individual results, exposure sources, and tailored strategies for exposure reduction. Participate in focus groups or interviews (subset only) to provide feedback on report clarity, usability, and communication preferences. This study focuses on rural adult residents of Nevada, including underserved populations who may face limited access to PFAS testing or environmental health education. Insights from this Phase I project will guide a future randomized controlled trial evaluating the intervention's broader impact on cardiovascular health and rural health equity.

DETAILED DESCRIPTION:
Background and Rationale: Per- and polyfluoroalkyl substances (PFAS) are a class of synthetic chemicals widely used in industrial and consumer products due to their water- and oil-repellent properties, as well as durability and resistance to heat. Because PFAS are highly persistent in the environment and human body, they are often referred to as "forever chemicals." PFAS are found in food packaging, non-stick cookware, stain- and water-resistant textiles, personal care products, carpets, and other household materials. Human exposure occurs primarily through contaminated drinking water, diet, consumer products, and inhalation of household dust. Nearly all individuals tested in the United States have measurable levels of PFAS in their blood. Chronic PFAS exposure has been linked to adverse health outcomes, including cardiometabolic disorders (hypertension, dyslipidemia, vascular disease, cardiac toxicity), endocrine and thyroid dysfunction, immune system impairment, congenital anomalies, liver disease, cancer, and developmental effects. Rural communities are disproportionately affected by PFAS exposure due to multiple factors, including reliance on small water utilities, private wells, proximity to industrial or military sites, and agricultural contamination from sludge-based fertilizers. These populations often face compounded health disparities, such as limited access to preventive healthcare, lower environmental health literacy (EHL), and higher baseline rates of chronic disease. National guidance, such as from the US National Academies of Sciences, Engineering, and Medicine (NASEM), recommends that individuals with elevated PFAS levels receive clinical monitoring for dyslipidemia and other health risks. However, rural residents and many healthcare providers lack practical, accessible tools to understand, interpret, and act upon PFAS exposure information. Previous research demonstrates that biomonitoring report-back-providing individuals with their personal chemical exposure results accompanied by actionable recommendations-can increase environmental health literacy, promote risk-reduction behaviors, and improve wellness outcomes without causing undue stress. Million Marker (MM), a direct-to-consumer biomonitoring company, has demonstrated success with report-back interventions for endocrine-disrupting chemicals (EDCs), showing improvements in EHL, behavior, and urinary biomarker levels. Leveraging this expertise, this study aims to develop and pilot an educational and actionable PFAS blood test report-back intervention for rural adults, in collaboration with healthcare providers, to improve knowledge, behavior, and wellness outcomes. Study Objectives: The primary goal of this observational study is to assess whether personalized PFAS blood test results combined with educational and actionable report-back materials can: 1. Increase environmental health literacy (EHL) regarding PFAS exposure and associated health risks. 2. Enhance readiness to reduce PFAS exposure and adoption of risk-reduction behaviors. 3. Improve wellness indicators, including stress reduction, sleep quality, and perceived control over health. Secondary objectives include evaluating usability and comprehension of the report-back materials, identifying barriers to behavioral change, and informing the design of a future Phase II randomized trial and scalable public health intervention. Study Design: This is a prospective, single-group observational study utilizing pre- and post-intervention surveys to evaluate outcomes. Participants will serve as their own control, with baseline measurements compared to post-intervention responses. The study incorporates both quantitative and qualitative methodologies to develop, refine, and evaluate the PFAS report-back intervention. Sample Size: The study will recruit 110 adult participants residing in rural areas. Sample size calculations, based on previous report-back interventions, ensure at least 80% power to detect meaningful changes in EHL and readiness to act, accounting for up to 16% attrition. Population and Eligibility: Inclusion criteria includes age ≥ 18 years, residing or working in a rural area of Nevada (verified via zip code and Health Resources and Services Administration classification), ability to understand English and complete study activities, and willingness to provide mail-in blood sample and complete pre- and post-surveys. Diversity and Representation: The study aims for at least 30% representation from minority populations, including Hispanic and Black residents, reflecting Nevada's rural demographics. Procedures: 1. Recruitment and Consent: Participants will be recruited via the Healthy Nevada Project, which maintains a population cohort of over 50,000 residents, including a substantial rural subset. Recruitment methods include targeted mailings and electronic communications. Interested participants will review study information and provide informed consent electronically. 2. Baseline Assessment: Participants will complete a pre-intervention survey capturing: demographics (age, gender, race/ethnicity, education, income), environmental health literacy (general and PFAS-specific knowledge, attitudes, and behaviors), lifestyle and exposure behaviors (diet, water use, product use, cleaning habits, and household exposures), and wellness measures (stress, sleep, and self-assessed health status). 3. PFAS Blood Sample Collection: Participants will receive a mail-in blood spot collection kit through Relentless Health. Instructions and a short video will guide participants through self-collection. Blood samples will be returned to the lab for PFAS biomarker analysis. 4. Report-Back Intervention: Each participant will receive a personalized PFAS report summarizing: individual PFAS biomarker concentrations, comparison with national reference data and NASEM guidance levels, identification of likely exposure sources, tailored, practical recommendations for reducing PFAS exposure (e.g., water filtration, product substitution, behavioral modifications), and suggestions for healthcare provider follow-up if results are above the 95th percentile. 5. Focus Groups and Interviews (Qualitative Component): A subset of participants (n≈20) and healthcare providers (n≈10) will engage in virtual focus groups or key informant interviews to provide feedback on report clarity, usability, and communication preferences. These sessions will inform iterative refinements to the report-back materials. 6. Post-Intervention Assessment: Two weeks after receiving their report, participants will complete a follow-up survey assessing: changes in PFAS-specific environmental health literacy, readiness and self-reported behaviors to reduce PFAS exposure, wellness outcomes (stress, sleep, empowerment), and usability, comprehension, and satisfaction with the report-back. Data Collection Instruments: PFAS Environmental Health Literacy Survey (developed and validated for this study), lifestyle and Exposure Audit (expanded to include PFAS-specific questions), and usability and Program Evaluation Questionnaire. Standardized wellness instruments: Perceived Stress Scale (PSS), Behavioral Risk Factor Surveillance System sleep and health modules, and Readiness to change survey based on the Transtheoretical Model of Health Behavior Change. Outcome Measures: Primary Outcomes: 1. Change in PFAS-specific environmental health literacy (pre- vs post-intervention), 2. Change in readiness to reduce PFAS exposure, 3. Change in wellness indicators (stress, sleep, perceived control). Secondary Outcomes: Usability, clarity, and satisfaction with the report-back materials, identification of barriers and facilitators to behavioral change, and qualitative themes on interpretation, comprehension, and behavioral intentions. Data Analysis Plan: Quantitative Analysis: Pre- and post-intervention outcomes will be compared using paired statistical tests (Student's t-test, Wilcoxon signed-rank test for non-normal distributions). Categorical variables will be assessed via chi-square tests. Reliability of PFAS-specific EHL survey will be evaluated using Cronbach's alpha. Secondary exploratory analyses will evaluate correlations between PFAS blood levels, EHL, and self-reported behavior change. Qualitative Analysis: Focus group and interview transcripts will be coded using NVivo software. Two independent coders will identify recurring themes; discrepancies will be resolved via discussion. Thematic analysis will inform report-back refinement, ensuring cultural relevance, clarity, and practicality for rural populations. Ethical Considerations: Participants will be informed of potential risks, including stress associated with receiving exposure results. Personalized counseling and guidance will be provided for individuals with elevated PFAS levels. Ethical principles of autonomy, beneficence, nonmaleficence, and justice will guide all study procedures. Gift card incentives will be provided for survey completion and focus group participation. Significance and Innovation: This study addresses rural health disparities by providing accessible PFAS testing and actionable educational interventions to populations at high risk of exposure. Innovations include: the first direct-to-consumer PFAS mail-in blood test with report-back designed for rural populations and healthcare providers, integration of PFAS biomonitoring with behavioral intervention principles grounded in Self-Regulation Theory, Self-Determination Theory, and the Theory of Planned Behavior, development of the first PFAS-specific environmental health literacy survey, and scalable, low-cost intervention potentially adaptable to other marginalized or underserved populations. Future Directions: Data generated in this Phase I study will inform a Phase II randomized controlled trial to evaluate long-term efficacy, cardiovascular health outcomes, and scalability. The intervention may ultimately be integrated into clinical care, public health programs, and broader population-level PFAS exposure mitigation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Residing or working in a rural area (verified via zip code and Health Resources and Services Administration classification)
* Ability to understand English and complete study activities
* Willingness to provide mail-in blood sample and complete pre- and post-surveys

Exclusion Criteria:

* Age<18
* Residing in an urban or suburban area
* Does not understand English or complete study activities
* Not willing to provide a mail-in blood sample and/or complete pre- and post- surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in PFAS Environmental Health Literacy | 4 weeks
  Change in PFAS-specific environmental health literacy (pre- vs post-intervention). Participants complete a 12 question survey with Likert type response options. Three subscales (4 questions each for knowledge, attitudes, and behavior) are summed separately, each with a minimum value of 4 and a maximum of 20. A higher score is considered better.
Change in response to a survey question assessing "Readiness to reduce PFAS exposure" | 4 weeks
  Participants are asked to choose the sentence (from among 5 options) that most accurately describes their current efforts and interest in limiting their exposure to PFAS. Each sentence reflects one of 5 stages of change, in order from earlier to later (better): precontemplation, contemplation, preparation, action, and maintenance. The post-intervention stage is compared to the pre-intervention stage to identify increased, decreased, or no change in readiness to reduce PFAS exposure after completing the intervention.

SECONDARY OUTCOMES:
Usability, clarity, and satisfaction with the report-back materials | 4 weeks
  This outcome uses the System Usability Scale, which is a series of 10 questions about usability of the report-back program, including clarity, ease of use and satisfaction. Responses are Likert style from Strongly disagree to Strongly Agree with 5 options ranging from 0 to 4. Direction varies with the questions and half are reverse coded in the scoring system, which results in a score between 0-100.
Identification of challenges to behavioral change | 4 weeks
  Participants are asked to identify whether each of nine questions naming possible challenges to reducing exposure to harmful chemicals is "true" for them, or "not true" for them. Each questions is evaluated individually, but described together as the percentage of participants choosing "true for me" for each question. Changes from pre- to post-intervention in the overall percentage for each question will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Kwiatkowski, Principal Investigator — Million Marker Wellness
Locations (1):
- Million Marker, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Million Marker will disseminate research results and findings to the scientific community through presentations at scientific meetings and conferences and publications in academic journals, as well as through the mass media and online postings. The Principal Investigator of this study will make data and associated documentation/metadata available to external researchers under a data-sharing agreement in which a specific commitment is made to use the data for research purposes only, to not provide the data to a third party or distribute it in any form, and to properly acknowledge the source of funding for the collection of the data and the researchers involved in this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: Researchers must submit an acceptable research plan (goals of the proposed research, the specific hypotheses to be examined, justification for research and methods), be affiliated with a recognized research institution, have demonstrated expertise in the area of the proposed research project, and receive independent approval from their governing institutional review board. Data will be available for use only to answer the specific question(s) indicated in the research plan. The researchers must provide a list of variable names and an outline of how research findings will be disseminated; and will be asked to sign a data-sharing agreement that commits to: 1) not attempt to identify any individual participant, 2) secure the data using appropriate software technology, 3) and destroy or return all data once analyses are complete. All final datasets will be de-identified. Final authorship on manuscripts will require review and approval by the Principal Investigators of this study.

REFERENCES:
- [Background] Carignan CC, Bauer RA, Patterson A, Phomsopha T, Redman E, Stapleton HM, Higgins CP. Self-Collection Blood Test for PFASs: Comparing Volumetric Microsamplers with a Traditional Serum Approach. Environ Sci Technol. 2023 May 30;57(21):7950-7957. doi: 10.1021/acs.est.2c09852. Epub 2023 May 15. PMID 37189231
- [Background] Rochester JR, Kwiatkowski CF, Neveux I, Dabe S, Hatcher KM, Lathrop MK, Daza EJ, Eskenazi B, Grzymski JJ, Hua J. A Personalized Intervention to Increase Environmental Health Literacy and Readiness to Change in a Northern Nevada Population: Effects of Environmental Chemical Exposure Report-Back. Int J Environ Res Public Health. 2024 Jul 11;21(7):905. doi: 10.3390/ijerph21070905. PMID 39063482
- [Background] Boronow KE, Cohn B, Havas L, Plumb M, Brody JG. The Effect of Individual or Study-Wide Report-Back on Knowledge, Concern, and Exposure-Reducing Behaviors Related to Endocrine-Disrupting Chemicals. Environ Health Perspect. 2023 Sep;131(9):97005. doi: 10.1289/EHP12565. Epub 2023 Sep 8. PMID 37682721
- [Background] Korfmacher KS, Brody JG. Moving Forward with Reporting Back Individual Environmental Health Research Results. Environ Health Perspect. 2023 Dec;131(12):125002. doi: 10.1289/EHP12463. Epub 2023 Dec 14. PMID 38095662
- [Background] Gehle KS, Crawford JL, Hatcher MT. Integrating environmental health into medical education. Am J Prev Med. 2011 Oct;41(4 Suppl 3):S296-301. doi: 10.1016/j.amepre.2011.06.007. PMID 21961679
- [Background] Finn S, O'Fallon L. The Emergence of Environmental Health Literacy-From Its Roots to Its Future Potential. Environ Health Perspect. 2017 Apr;125(4):495-501. doi: 10.1289/ehp.1409337. Epub 2015 Jun 30. PMID 26126293
- [Background] Johnston J, Cushing L. Chemical Exposures, Health, and Environmental Justice in Communities Living on the Fenceline of Industry. Curr Environ Health Rep. 2020 Mar;7(1):48-57. doi: 10.1007/s40572-020-00263-8. PMID 31970715
- [Background] Bullard RD, Wright BH. Environmental justice for all: community perspectives on health and research needs. Toxicol Ind Health. 1993 Sep-Oct;9(5):821-41. doi: 10.1177/074823379300900508. PMID 8184445
- [Background] Hill-Briggs F, Ephraim PL, Vrany EA, Davidson KW, Pekmezaris R, Salas-Lopez D, Alfano CM, Gary-Webb TL. Social Determinants of Health, Race, and Diabetes Population Health Improvement: Black/African Americans as a Population Exemplar. Curr Diab Rep. 2022 Mar;22(3):117-128. doi: 10.1007/s11892-022-01454-3. Epub 2022 Mar 3. PMID 35239086
- [Background] United States Environmental Protection Agency. Biden-Harris Administration Finalizes First-Ever National Drinking Water Standard to Protect 100M People from PFAS Pollution. https://www.epa.gov/newsreleases/biden-harris-administration-finalizes-first-ever-national-drinking-water-standard (accessed 2024-06-05).
- [Background] C8 Science Panel. C8 Probable Link Reports. C8 Science Panel. http://c8sciencepanel.org/prob_link.html (accessed 2024-06-05).
- [Background] Fenton SE, Ducatman A, Boobis A, DeWitt JC, Lau C, Ng C, Smith JS, Roberts SM. Per- and Polyfluoroalkyl Substance Toxicity and Human Health Review: Current State of Knowledge and Strategies for Informing Future Research. Environ Toxicol Chem. 2021 Mar;40(3):606-630. doi: 10.1002/etc.4890. Epub 2020 Dec 7. PMID 33017053
- [Background] Blake BE, Fenton SE. Early life exposure to per- and polyfluoroalkyl substances (PFAS) and latent health outcomes: A review including the placenta as a target tissue and possible driver of peri- and postnatal effects. Toxicology. 2020 Oct;443:152565. doi: 10.1016/j.tox.2020.152565. Epub 2020 Aug 27. PMID 32861749
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Division on Earth and Life Studies; Board on Population Health and Public Health Practice; Board on Environmental Studies and Toxicology; Committee on the Guidance on PFAS Testing and Health Outcomes. Guidance on PFAS Exposure, Testing, and Clinical Follow-Up. Washington (DC): National Academies Press (US); 2022 Jul 28. Available from http://www.ncbi.nlm.nih.gov/books/NBK582439/ PMID 35939564
- [Background] Wen ZJ, Wei YJ, Zhang YF, Zhang YF. A review of cardiovascular effects and underlying mechanisms of legacy and emerging per- and polyfluoroalkyl substances (PFAS). Arch Toxicol. 2023 May;97(5):1195-1245. doi: 10.1007/s00204-023-03477-5. Epub 2023 Mar 22. PMID 36947184
- [Background] Liang Y, Zhou H, Zhang J, Li S, Shen W, Lei L. Exposure to perfluoroalkyl and polyfluoroalkyl substances and estimated glomerular filtration rate in adults: a cross-sectional study based on NHANES (2017-2018). Environ Sci Pollut Res Int. 2023 Apr;30(20):57931-57944. doi: 10.1007/s11356-023-26384-9. Epub 2023 Mar 27. PMID 36971931
- [Background] Sunderland EM, Hu XC, Dassuncao C, Tokranov AK, Wagner CC, Allen JG. A review of the pathways of human exposure to poly- and perfluoroalkyl substances (PFASs) and present understanding of health effects. J Expo Sci Environ Epidemiol. 2019 Mar;29(2):131-147. doi: 10.1038/s41370-018-0094-1. Epub 2018 Nov 23. PMID 30470793
- [Background] Cousins IT, Johansson JH, Salter ME, Sha B, Scheringer M. Outside the Safe Operating Space of a New Planetary Boundary for Per- and Polyfluoroalkyl Substances (PFAS). Environ Sci Technol. 2022 Aug 16;56(16):11172-11179. doi: 10.1021/acs.est.2c02765. Epub 2022 Aug 2. PMID 35916421
- [Background] Gluge J , Scheringer M , Cousins IT , DeWitt JC , Goldenman G , Herzke D , Lohmann R , Ng CA , Trier X , Wang Z . An overview of the uses of per- and polyfluoroalkyl substances (PFAS). Environ Sci Process Impacts. 2020 Dec 1;22(12):2345-2373. doi: 10.1039/d0em00291g. Epub 2020 Oct 30. PMID 33125022